CLINICAL TRIAL: NCT00442520
Title: Pharmacogenomic Study in Patients of Lung, Colorectal and Head/Neck Cancers Receiving Chemotherapy
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Paul J. Patton Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: 10270
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Lung Cancer; Colorectal Cancer; Head and Neck Cancer
MeSH Terms: conditions — Lung Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 2: colorectal cancer patients
- 3: head and neck cancer patients
- 1: lung cancer patients

SUMMARY:
The purpose of this study is to look at several genes that might determine how the body processes the drugs used to treat lung, colorectal and head and neck cancers. The goal of this examination is to help investigators determine the proper dosage to give future cancer patients or to better predict which future patients will respond to particular drug therapies.

DETAILED DESCRIPTION:
This study is to establish a pilot pharmacogenomic program in identifying genetic variation to predict the safety, toxicity and/or efficacy of drugs. DNA will be extracted from patients' peripheral blood to study SNPs in DPD, TS, MTHFR, UGT1A1, CYP3A4, CYP3A5, GSTM1, GSTT1, GSTP1, HO-1, ERCC1, XPD, XRCC1 and EGFR genes. The results of genetic study will be compared to treatment efficacy and toxicity. The ultimate goal is to use genotype profiles to provide individualized cancer treatment to improve outcome and decrease toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Lung, Colorectal and Head and Neck Cancer Patients that have received or plan to receive chemotherapy as part of their treatment

Exclusion Criteria:

* Colorectal cancer patients that have never received or will not receive chemotherapy as part of their therapy
* Head and Neck cancer patients that have never received or will not receive chemotherapy as part of their treatment
* Patients with cancer types other than colorectal or head and neck
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: medical center
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2006-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Jui Yvonne Wan, Ph.D., Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States